CLINICAL TRIAL: NCT04307082
Title: A Phase 1, Open-Label, Single-Centre Study to Evaluate the Absorption, Distribution, Metabolism, and Excretion (ADME) of Oral [14C]-Ibrexafungerp in Healthy Male Subjects
Brief Title: ADME Study of [14C]-Ibrexafungerp in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Scynexis, Inc. (Industry)
Collaborators: Inncelerex (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SCY-078-116
Record Dates: First submitted 2020-03-04; First posted 2020-03-13 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Fungal Infection
Keywords: SCY-078; Ibrexafungerp; ADME
MeSH Terms: conditions — Mycoses

STUDY DESIGN:
Intervention Model Description: Open Label, single arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ibrexafungerp (Experimental): Oral [14C]-Ibrexafungerp Single Dose
  Interventions: Drug: [14C]-Ibrexafungerp

INTERVENTIONS:
Drug: [14C]-Ibrexafungerp — Radio-labeled Ibrexafungerp, single dose.
  Other Names: [14C]-SCY-078

SUMMARY:
This is a Phase 1, open-label, single-centre, non-randomised study to evaluate the absorption, distribution, metabolism, and excretion (ADME) of an oral solution of [14C]-ibrexafungerp following administration in healthy male subjects.

Each subject will receive a single dose of [14C]-ibrexafungerp and will be followed for up to 20 days. During this period total radioactivity will be measured in blood, urine and faeces.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, single-centre, non-randomised study to evaluate the absorption, distribution, metabolism, and excretion (ADME) of an oral solution of [14C]-ibrexafungerp following administration in healthy male subjects.

Each subject will receive a single dose of [14C]-ibrexafungerp and will be followed for up to 20 days. During this period total radioactivity will be measured in blood, urine and faeces.

All subjects will undergo preliminary screening procedures for the study at the screening visit. Subjects will be admitted to the clinical unit on the evening prior to dosing (Day -1). A single oral dose containing [14C]-ibrexafungerp oral solution will be administered to subjects. Individual subjects will be released from the clinical unit following study-related procedures on Days 8 to 20 according to their % of radioactivity collected in relation to the dose administered.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy males
* Age 30 to 65 years of age at the time of signing informed consent
* Must be willing and able to participate in the whole study
* Must provide written informed consent
* Must agree to adhere to the contraception requirements

Key Exclusion Criteria:

* Subjects who have received any investigational drug in a clinical research study within the 90 days prior to Day 1
* Current smokers
* Recent radiation exposure
* Subjects who have been enrolled in a 14C ADME study in the last 12 months
* An acute or chronic disease determined by the investigator to be clinically significant
* Clinically significant abnormal clinical chemistry, haematology, coagulation or urinalysis at screening as judged by the investigator
* Evidence of renal impairment at screening
* History of clinically significant cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal disease, neurological or psychiatric disorder

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Mass balance | Day 20
  Amount recovered expressed as a percentage of the dose administered

SECONDARY OUTCOMES:
Routes and rates of elimination of [14C]-ibrexafungerp | Day 20
  Metabolite concentrations in body fluids and excreta
Number of subjects with treatment-emergent adverse events | Day 20
  Number of subjects with treatment-emergent adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Nkechi Azie, MD, Study Director — Scynexis, Inc.
Locations (1):
- Quotient Sciences, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No